## Appendix B: Participant consent form

Related to 'Nutrition and Pregnancy'

- I have read the information letter. I could also ask questions. My questions have been answered correctly. I had enough time to decide whether to participate.
- I know that participation is voluntary. I also know that I can decide at any time not to participate in the study. Or to stop. Then I don't have to say why I want to stop.
- I give the researchers permission to collect and use my data. The researchers only do this to answer the research question of this study.
- I know some people can view all my data to check the research. These people are listed in this information letter. I give these people permission to view my data for this check

| check. | | |
|---|---|---|
| <ul> <li>Would you like to tick yes or no below?</li> <li>I give permission to be asked after this study whether I would lik participate in a follow-up study.</li> </ul> | e to | Yes □ |
| - I want to participate in this study. | | |
| My name is (subject): | | |
| Signature: | Date :/ | / |
| I declare that I have fully informed this subject about the said research. | | |
| Name of the researcher (or his representative): | | |
| Signature: | Date: / / _ | _ |
| <if applicable=""></if> | | |
| Additional information has been provided by: Name: | | |
| Function: | | |

The subject will receive a complete information letter, together with a signed version of the consent form.

Signature:....

Date: \_\_ / \_\_ / \_\_

No□